CLINICAL TRIAL: NCT00148486
Title: A Fourteen-week Placebo-controlled Dose-response Efficacy and Safety Study of NS 2330 in Early Parkinson's Disease Patients (Study for Proof of Concept in Early Parkinson's Disease of a Triple Reuptake Inhibitor, NS 2330 / SCEPTRE)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1198.100
Record Dates: First submitted 2005-09-07; First posted 2005-09-08 (Estimated); Last update posted 2013-10-29 (Estimated); Status verified 2013-10

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Tesofensine

INTERVENTIONS:
Drug: NS 2330

SUMMARY:
To demonstrate efficacy and dose-response of NS 2330 versus placebo in patients with early Parkinson's Disease in 14 weeks of treatment, and to investigate the safety and tolerability of NS 2330 in these patients.

ELIGIBILITY:
Parkinson's disease for <5 years, non-demented, no or <6 months of levodopa and none during trial. Off levodopa, DA agonists, and psychotropics for 30 days before screening. Amantadine, anticholinergics allowed if at stable dosage. Hoehn & Yahr stage I-III. Depression allowed, but no other chronic disease that is unstable or might interfere with ability to participate.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 261
Dates: Start 2003-06; Primary Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
Mean change from Baseline to Week 14 in the score of the UPDRS, Parts I-III combined | baseline and 14 Weeks
Proportion of patients who were withdrawn from the study due to AEs | baseline and 14 Weeks

SECONDARY OUTCOMES:
Mean change in Part I, Part II, and Part III (separately) of the UPDRS | 14 weeks
Mean change in the Clinical Global Impressions (CGI)-Severity scale | 14 weeks
Mean change in the Modified Hoehn and Yahr Scale (MHYS) | 14 weeks
Mean change in the Modified Schwab-England Disability Scale (MSED) | 14 weeks
Mean change in the Hamilton Depression Scale (HAMD) (GRID version) (including an additional analysis of the subset of patients with a pretreatment [screening] score of 14 or more) | 14 weeks
Mean change in Snaith-Hamilton Pleasure Scale (SHAPS) (including an additional analysis of the subset of patients with a pretreatment [screening] score of 3 or more) | 14 weeks
Mean change in the Auditory Verbal Learning Test (AVLT) | 14 weeks
mean score at Week 14 on the CGI-Improvement (which has no baseline rating) | 14 weeks
Proportion of responder patients (20% and 30% improved on the total score of the UPDRS) | 14 weeks
Incidence of adverse events | 2 weeks
vital signs (blood pressure and pulse rate) | 20 weeks
patients with abnormal laboratory test measurements | 20 weeks
patients with abnormalities in electrocardiograms (ECGs) | 20 weeks
Epworth Sleepiness Scale (ESS) (for daytime sleepiness) | 20 weeks
Pittsburgh Sleep Quality Index (PSQI) for quality and pattern of sleep | 20 weeks
Drug plasma concentration | 20 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim Study Coordinator, Study Chair — Boehringer Ingelheim
Locations (55):
- United States (47):
  - Pivotal Reaserch Centers, Peoria, Arizona
  - Boehringer Ingelheim Investigational Site, Tucson, Arizona
  - PMDI, Fountain Valley, California
  - Boehringer Ingelheim Investigational Site, Fresno, California
  - Boehringer Ingelheim Investigational Site, Irvine, California
  - Boehringer Ingelheim Investigational Site, Ocenside, California
  - Boehringer Ingelheim Investigational Site, Oxnard, California
  - West Los Angeles VA Medical Center, West Los Angeles, California
  - Boehringer Ingelheim Investigational Site, Danbury, Connecticut
  - UCONN Health Center, Farmington, Connecticut
  - 60 Temple St, New Haven, Connecticut
  - Boehringer Ingelheim Investigational Site, Boca Raton, Florida
  - Boehringer Ingelheim Investigational Site, Bradenton, Florida
  - University of Florida, Gainsville, Florida
  - Sunrise Clinical Research, Hollywood, Florida
  - Department of Neurology, Miami, Florida
  - Miami Research Associates, Miami, Florida
  - Boehringer Ingelheim Investigational Site, Ocala, Florida
  - Renstar Medical Research, Ocala, Florida
  - Boehringer Ingelheim Investigational Site, Panama City, Florida
  - CNS Clinical Trials, Saint Piresburg, Florida
  - Movement Disorder Center, Tampa, Florida
  - University of Southern Florida, Tampa, Florida
  - Department of Neurological Sciences, Chicago, Illinois
  - Boehringer Ingelheim Investigational Site, Fort Wayne, Indiana
  - Outpatient Clinical Research Facility, Indianapolis, Indiana
  - Boehringer Ingelheim Investigational Site, Kansas City, Kansas
  - Boehringer Ingelheim Investigational Site, Shreveport, Louisiana
  - Boehringer Ingelheim Investigational Site, Scarborough, Maine
  - Boehringer Ingelheim Investigational Site, Springfield, Massachusetts
  - Future Care Studies, Springfield, Massachusetts
  - Boehringer Ingelheim Investigational Site, Traverse City, Michigan
  - Boehringer Ingelheim Investigational Site, Minneapolis, Minnesota
  - University of Minesota, Minneapolis, Minnesota
  - Boehringer Ingelheim Investigational Site, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Global Medical Institutes LLC, Toms River, New Jersey
  - Upstate Clinical Resaerch LLC, Albany, New York
  - Boehringer Ingelheim Investigational Site, New York, New York
  - Boehringer Ingelheim Investigational Site, Wiston-Salem, North Carolina
  - Ohio State University Medical Center, Columbus, Ohio
  - Neurology Specialists Inc., Dayton, Ohio
  - St. John's Doctor Building, Tulsa, Oklahoma
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - The Methodist Hospital, Houston, Texas
  - Boehringer Ingelheim Investigational Site, San Antonio, Texas
  - North Texas Neurology Associates, Wichita Falls, Texas
- Canada (8):
  - University of Calgary, Calgary, Alberta
  - University of British Columbia, Vancouver, British Columbia
  - Davidson Memory Clinic, Moncton, New Brunswick
  - Boehringer Ingelheim Investigational Site, Halifax, Nova Scotia
  - Centre For Movement Disorders, Markham, Ontario
  - Clinical Research Consultant Group, Beaconsfield, Quebec
  - Memory and Motor Skills Disorders Clinic, Québec, Quebec
  - Boehringer Ingelheim Investigational Site, Saskatoon, Saskatchewan